CLINICAL TRIAL: NCT06286345
Title: Lifestyle InterVEntion Study in General Practice: LIVES - GP
Acronym: LIVES-GP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: GGZ Drenthe Mental Health Institution (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17644
Record Dates: First submitted 2024-02-05; First posted 2024-02-29 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Depression, Unipolar; Cardiovascular Diseases
Keywords: depression; lifestyle; general practice
MeSH Terms: conditions — Depressive Disorder; Cardiovascular Diseases; Depression

STUDY DESIGN:
Intervention Model Description: Uncontrolled cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: GLI-LEEF — GLI-LEEF is an 18-week program, during which various lifestyle topics are discussed, such as nutrition, exercise, sleep, relationships and intimacy, and specific education about depression and its influence on lifestyle. GLI-LEEF is aimed at improving the activity level, quality of life and (cardiovascular) health of patients and thus increasing the general functioning and well-being of patients and at the same time reducing psychological complaints.
  GLI-LEEF consists of 14 group meetings and 4 individual meetings, the group meetings last 90 minutes, the individual meetings 30 minutes. Patients are asked to wear a FitBit and to complete short homework assignments. Each group contains 8-10 patients. Patients are asked to find a buddy who can support them during the program.

SUMMARY:
Patients with depression are at a substantially increased risk of chronic physical disease including cardiovascular disease. This may be attributed primarily to an unhealthy lifestyle related to their disorder. Interestingly, the unhealthy lifestyle feeds back to decreased quality of life and increased depressive symptoms, thus creating a hazardous vicious circle. Consequently, there is a great potential for 'Lifestyle Medicine' for depression. Yet, it is known that patients with depression often have motivational and self-management problems. Therefore an 18 session multimodal lifestyle intervention (MLI) specifically tailored to the needs of depressed patients was developed and piloted in mental health care, with promising results. This research aims to investigate using a process evaluation the feasibility of this MLI in general practice because this is the setting where the majority of patients with depression are treated and results from mental health care are unlikely to apply.

DETAILED DESCRIPTION:
Rationale: Patients with depression are at a substantially increased risk of chronic physical disease including cardiovascular disease. This may be attributed primarily to an unhealthy lifestyle related to their disorder. Interestingly, the unhealthy lifestyle feeds back to decreased quality of life and increased depressive symptoms, thus creating a hazardous vicious circle. Consequently, there is a great potential for 'Lifestyle Medicine' for depression. Yet, it is known that patients with depression often have motivational and self-management problems. Therefore a multimodal lifestyle intervention (MLI) specifically tailored to the needs of depressed patients was developed and piloted in mental health care, with promising results. This research aims to investigate this MLI in general practice because this is the setting where the majority of patients with depression are treated and results from mental health care are unlikely to apply.

Objective: to estimate in general practice the feasibility of conducting a large-scale study on the effectiveness of a MLI for depression, and identify key factors that can influence its successful conduct. In addition, this study aims to obtain an estimate of the variance of outcome measures (mental health, lifestyle factors, functioning, recovery, wellbeing, sleeping quality, self-esteem, quality of life, health care costs, anthropometry and blood pressure).

Study design: An observational single-group prospective cohort study (n = 50) using mixed methods with baseline measurement and two follow-up measurements: after the intervention at 18 weeks and after a follow-up at 42 weeks.

Study population: Patients (18 years or over) with depression and overweight who are being treated in general practice.

Intervention (if applicable): A MLI named (in Dutch) "Gecombineerde Leefstijl Interventie Leef" (GLI-LEEF), developed for patients with depression consisting of several modules (e.g. on physical activity, healthy diet) comprising both individual and group sessions.

Main study parameters/endpoints: implementation feasibility using three of the elements of the 'Reach, Effectiveness, Adoption, Implementation, Maintenance' (RE-AIM) framework for process evaluation (i.e. Reach, Adoption and Implementation)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depressive symptoms or depressive disorder in the past year as registered in the general practice electronic health record and coded according to the International Classification of Primary Care (ICPC) as P03 and P76, respectively, or currently treated for depressive symptoms or depressive disorder in general practice.
* At least mild depressive symptom level according to the Quick Inventory Depressive Symptomatology-Self-Report (QIDS-SR) (score ≥6)
* Body mass index ≥ 25 kg/m2 or increased waist circumference (>88 cm (women) of >102 cm (men)).

Exclusion Criteria:

* Current treatment in mental health care (GGZ in Dutch)
* Severe somatic / neurological disease at the discretion of the GP
* Currently participating in another lifestyle intervention
* Insufficient proficiency in Dutch
* Inability to read and write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Reach of GLI-LEEF | 12 months
  Reach of GLI-LEEF as defined as the number of individuals who are willing to participate in this study
General practice adoption of GLI-LEEF | 12 months
  General practice adoption of GLI-LEEF as defined by the number of general practices that are willing to implement GLI-LEEF in this study
General practitioner adoption of GLI-LEEF | 12 months
  General practice adoption of GLI-LEEF as defined by the number of general practitioners that are willing to implement GLI-LEEF in this study
Lifestyle coach adoption of GLI-LEEF | 12 months
  Lifestyle coach adoption of GLI-LEEF as defined by the number of lifestyle coaches that are willing to implement GLI-LEEF in this study
Adherence to GLI-LEEF | 18 weeks
  First aspect of implementation is adherence to GLI-LEEF which is defined by the number of sessions attended by the participant out of the total of 18 sessions
Drop-out from GLI-LEEF | 18 weeks
  Second aspect of implementation is drop-out from GLI-LEEF which is defined by the proportion of participants who decide to prematurely stop taking part in the intervention
Barriers and facilitators of the GLI-LEEF implementation | 18 weeks
  Potential barriers and facilitators of the GLI-LEEF implementation will be identified using a qualitative approach by interviewing approximately 10 participants who dropped out and 10 who completed GLI-LEEF, if opportune

SECONDARY OUTCOMES:
Body weight of the participant as assessed by a medical weight scale | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  Body weight in kilograms
Body height of the participant as assessed by a stadiometer | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  Body height in meters
Waist circumference of the participant as assessed using a tape meter line | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  Waist circumference in centimeters
Diastolic and systolic blood pressure as assessed using a sphygmomanometer | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  Diastolic and systolic blood pressure in millimeters mercury
Treatment success on several domains by according to the Outcome Questionnaire-45 (OQ-=45) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The OQ-45 runs from 0 to 180. The lower the score, the more successful treatment
Recovery of the participant according to the Individual Recovery Outcomes - Counter (I.ROC) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The I.ROC is an instrument to quantitatively measure recovery. The total score runs from 12 to 72. Higher scores indicate better outcomes.
Wellbeing as assessed by the Mental Health Continuum Short Form (MHC-SF) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The MHC-SF measures emotional, social and psychological wellbeing. Its total score runs from 0 to 20. Higher score means better outcome.
Self esteem according to the Rosenberg Self-Esteem Scale (RSES) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The RSES is a widely used self-report instrument for evaluating individual self-esteem. The total score runs from 0 to 30. Higher score means worse outcome, i.e. less self-esteem.
Insomnia according to the Insomnia Severity Index (ISI) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The ISI assesses insomnia. The total score runs from 0 to 28. Higher score means worse outcome.
Quality of life according to the Recovering Quality of Life (ReQol) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  This is a Patient Reported Outcome Measure assesses the quality of life for people with different mental health conditions. Its score runs from 0 to 80. Higher score means better outcome.
Health care consumption and productivity loss according to the Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P) | Baseline, at the end of the intervention (18 weeks), and at the 6 months follow up (42 weeks after baseline)
  The TiC - P assesses health care consumption and productivity loss in patients with mental illness

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands